CLINICAL TRIAL: NCT02278627
Title: Impact of a Technique of Massage During the First Week of Hospitalization on the Recycling of the Mobility of the Knee Further to the Installation of Knee Replacement
Acronym: PTGMass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: I11002
Record Dates: First submitted 2014-09-11; First posted 2014-10-30 (Estimated); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Orthopedic Surgery
MeSH Terms: interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- manual lymphatic drainage (Experimental): We wish to complete the physiotherapist's support with manual lymphatic drainage (MLD) using a specific method based on pressure of finger splayed (PFS)
  Interventions: Other: manual lymphatic drainage
- Usual treatment (No Intervention)

INTERVENTIONS:
Other: manual lymphatic drainage
  Arms: manual lymphatic drainage

SUMMARY:
During fthe first postoperative days, physiotherapists supported patients with knee replacement in orthopaedics of Saint-Junien's and Limoges' hospitals. This support includes movements of the leg in active and non active motions, without any help and with an arthromotor, and involves walking rehabilitation.

The investigators would like to complete the physiotherapist's support with manual lymphatic drainage (MLD) using a specific method based on pressure of finger splayed (PFS). This might have a positive impact on time recovery of joint range, on postoperative oedema resorbtion and on patient's pain during rehabilitation classes.

French National Authority for Health specifies there is not a single study assessing massage effects on knee replacement, according to current bibliography.

The investigators purpose is the establishment of a prospective, controlled, randomised trial referred as a "superiority" trial. A total of 98 patients divided in 2 parallel groups will be created.

The study will be in an open-label manner for both patient and physiotherapist involved in walk rehabilitation but will be conducted as a blinded study for the investigating physiotherapist.

Inclusion period will be 17 months and the following period will be 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* At least 18-years-old patients.
* Men and women operated for a knee replacement.
* Patients affiliated to a social security system and having given their informed consent write.

Exclusion Criteria:

* Patients operated on Fridays
* Patients presenting contraindications to the administration of a treatment by héparine
* Patients affected by insane pathology or by confusion.
* Patients participating in another medical research
* Pregnant and breast-feeding women and without effective contraception.
* Patients under guardianship or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-09; Primary Completion 2017-04 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
To measure the joint range at day 7 after operation | 2 days (Day 0 and Day 7)
  The measures will be made with a goniometer

SECONDARY OUTCOMES:
To measure the oedema at day 7 after operation | 2 days (Day 0 and Day 7)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Limoges, Limoges, France